CLINICAL TRIAL: NCT05213013
Title: The Effect of Toy-Type Nebulizer on Fear and Anxiety in Children Receiving Inhaler Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aylin Kurt (Other)
Responsible Party: Sponsor-Investigator, Aylin Kurt, Principal Investigator, Bartın Unıversity
Organization: Bartın Unıversity (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2021-SBB-0333
Record Dates: First submitted 2021-12-04; First posted 2022-01-28 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Children, Only; Fear Anxiety; Hospitalism in Children

STUDY DESIGN:
Intervention Model Description: Children and their parents
Who Masked: Participant, Care Provider
Masking Description: Children and their parents
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): All registered participants in the control group, will receive inhaler treatment with the toy-type nebulizer in the hospital. Both the parent and the child in the intervention group will be trained on the use of a nebulizer/mask.
  Interventions: Other: inhaler treatment with the toy-type nebulizer and training on on the use of a nebulizer/mask
- No intervention (No Intervention): No intervention. All registered participants in the control group, will receive inhaler treatment with the standard nebulizer in the hospital. Both the parent and the child in the intervention group will not be trained on the use of a nebulizer/mask.

INTERVENTIONS:
Other: inhaler treatment with the toy-type nebulizer and training on on the use of a nebulizer/mask — The children (experimental group), will receive training and inhaler treatment with the toy-type nebulizer. The training topics is as follows:
  * For effective nebulization, it should be ensured that the parts of the mask are assembled completely and correctly.
  * The child should be in an upright sitting position during nebulization.
  * During the procedure, normal breathing should be given into the mask.
  * As the medicine is finished, a sizzling sound is heard from the device.
  * After the nebula is over, the face should be washed and the mouth should be rinsed to remove the drug residues accumulated on the face and mouth.
  Arms: Experimental

SUMMARY:
The aim of this study is to determine the effect of toy-type nebulizers on fear and anxiety in children receiving inhaler therapy.

The research hypotheses are as follows:

H0: There is no significant difference between the intervention group and the the control group in the mean score of the "Child Fear Scale" and "Child Anxiety Scale-State" during and after the inhaler treatment with a toy-type nebulizer. H1: During and after the s inhaler treatment with the toy-type nebulizer, the mean score of the "Child Fear Scale" and "Child Anxiety Scale-State" is significantly higher in the intervention group compared to the control group.

DETAILED DESCRIPTION:
In this study, there will be two groups as the intervention (who will receive inhaler treatment with an education and toy type nebulizer) and the control group (who will not receive training and will receive inhaler treatment with a classic-looking nebulizer). A power analysis was performed based on the number of children in both groups, based on another study using the scales to be used in the research. According to the calculations made in the G-Power 3.1 Demo package program, when the effect size was accepted as 0.8, it was seen that at least 32 cases in each group would be sufficient for 80% power. Children who meet the research criteria will be randomly assigned to the intervention and control groups via http://www.randomize.org/ by assigning a number to the order of arrival at the hospital.

Inhaler treatment will be applied to both the intervention and control groups. Both the parent and the child in the intervention group will be trained on the use of a nebulizer/mask. The children in the intervention group will be treated with a toy-type nebulizer and the group will be treated with an inhaler, and the control group will be given inhaler treatment with the standard nebulizer in the hospital. Two researchers were employed for the inhaler treatment both for the intervention and control groups. One researcher performed the inhaler treatment for all children and the other researcher helped the children to assess their fear and anxiety level. Fear and anxiety in children were evaluated by the children and their parents who before, during, and the procedure, and five minutes after the procedure. The inhaler treatment procedure was performed by the same researcher both in the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* The child is between the ages of 4-10
* The child's application to the Pediatric Emergency Unit
* Child receiving inhaler treatment for the first time
* Parent and child agreeing to participate in the project
* Absence of speech and visual impairment of the child and his parents

Exclusion Criteria:

* The child is not between the ages of 4-10
* The child's application to another department except for the Pediatric Emergency Unit
* Child not receiving inhaler treatment for the first time
* Parent and child not agreeing to participate in the project
* Having speech and visual impairment of the child and his parents

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2022-01-30 (Actual); Primary Completion 2023-01-28 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Difference between the mean score of the "Child Fear Scale" between intervention and control groups | 12 months
  "The Child Fear Scale" will be completed before training and inhaler treatment with toy-type treatment that gathers quantitative data that will fear about the inhaler treatment with a nebulizer in children. This scale will also be completed at the intervention during and ten minutes after the intervention. The quantitative data will be used to measure a change in the children's fear level before, during and after the proposed intervention. The scale will be made without training and inhaler treatment with a standard nebulizer in the control group. At the end of the study, difference between the mean score of "The Child Fear Scale" between intervention and control groups will be examined. The Child Fear Scale total score mean of the children in the intervention group will be higher after the intervention compared to the control group. Data will be analyzed using Statistical Package for the Social Sciences package program.
Difference between the mean score of "The Child Anxiety Meter-State" between intervention and control groups | 12 months
  "The Child Anxiety Meter-State" will be completed before training and inhaler treatment with toy-type treatment that gathers quantitative data that will anxiety about the inhaler treatment with a nebulizer in children. This scale will also be completed at the intervention during and ten minutes after the intervention. The quantitative data will be used to measure a change in the children's anxiety level before, during and after the proposed intervention. The scale will be made without training and inhaler treatment with a standard nebulizer in the control group. At the end of the study, difference between the mean score of "The Child Anxiety Meter-State" between intervention and control groups will be examined. The Child Anxiety Meter-State total score mean of the children in the intervention group will be higher after the intervention compared to the control group. Data will be analyzed using Statistical Package for the Social Sciences package program.

SECONDARY OUTCOMES:
Change of the mean scores obtained by the children in the intervention group from the "Child Fear Scale" before and after the intervention. | 12 months
  "The Child Fear Scale" will be completed before training and inhaler treatment with toy-type treatment that gathers quantitative data that will address fear about the inhaler treatment with a nebulizer in children. These surveys will also be completed at the intervention during and ten minutes after the intervention. The quantitative data will be used to measure a change in the children's fear before, during and after the proposed intervention. The Child Fear Scale total score mean of the children in the intervention group will be higher after the intervention. Data will be analyzed using Statistical Package for the Social Sciences package program.
Change of the mean scores obtained by the children in the intervention group from the "Child Anxiety Meter-State" before and after the intervention. | 12 months
  "The Child Anxiety Meter-State" will be completed before training and inhaler treatment with toy-type treatment that gathers quantitative data that will address anxiety about the inhaler treatment with a nebulizer in children. These surveys will also be completed at the intervention during and ten minutes after the intervention. The quantitative data will be used to measure a change in the children's anxiety before, during and after the proposed intervention. The Child Anxiety Meter-State total score mean of the children in the intervention group will be higher after the intervention. Data will be analyzed using Statistical Package for the Social Sciences package program.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 12 months